CLINICAL TRIAL: NCT01190592
Title: Effects of Resistance Training With Milk Supplementation on Body Composition in Middle School Children
Brief Title: Resistance Training With Milk Supplementation in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Joesph E. Donnelly & Richard Washburn, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11935; NCT01787734 (obsolete NCT alias)
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Body Composition; Cardiovascular Risk Factors
Keywords: Resistance training; Body Composition; Cardiovascular Risk factors; Dairy
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Milk (Experimental)
  Interventions: Other: Resistance Training with Milk Supplementation in Adolescents
- Juice (Experimental)
  Interventions: Other: Resistance Training with Milk Supplementation in Adolescents
- Water (Placebo Comparator)
  Interventions: Other: Resistance Training with Milk Supplementation in Adolescents

INTERVENTIONS:
Other: Resistance Training with Milk Supplementation in Adolescents — On resistance training days, the RT+ milk group will receive milk (280kcals) immediately following exercise and milk at another time during the day. The RT+ juice group will receive fruit juice immediately following resistance exercise and juice again another time during the day. The RT+ water group will receive water following resistance exercise and water at another time during the day.
  On non training days, students in the RT+ milk group will receive milk. Students in the RT+ juice group will receive juice. The RT+ water group will receive water during the school day. On non-RT days, the total volume of milk, juice, or water will be split into two administration times during the school day.

SUMMARY:
The investigators primary objective is to evaluate the effect of a 6 month (3 days/wk) supervised, progressive RT program with increased daily milk intake in untrained adolescents on measures of body composition and cardiovascular risk factors. The investigators hypothesize that milk supplementation will produce significantly greater favorable changes in all body composition measures compared with RT + carbohydrate and control.

DETAILED DESCRIPTION:
We will recruit 150 healthy, adolescent middle school boys and girls (grades 7 through 9), BMI > 50th percentile < 98th percentile, who will participate in 6 months of supervised resistance training (3 days/wk) and will be randomized to one of 3 groups: RT + milk, RT + isocaloric carbohydrate, RT only (control). Both physical activity and diet outside the study protocol will be carefully monitored. Measurements will be completed at baseline 3 months and upon completion of the training protocol at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Middle school student (Grades 7-9)
2. BMI > 50th percentile - < 98th percentile
3. No resistance training in the past 6 months.
4. Endurance training (running, cycling, swimming, walking for exercise etc) not more than 3 hr per week, as assessed by screening questionnaire.
5. Weight stable (+/- 4.5kg) for 3 months prior to intake.
6. Willing to be randomized to one of the 3 study groups.

Exclusion criteria:

1. Individuals with contraindications based on review of health history by the investigators, including blood pressure, lipid profile, glucose, and insulin, and abnormal values obtained in a 24 item blood panel, such as electrolytes, liver function, etc. These individuals will be referred to their primary care physician for further evaluation and to obtain permission to participate. The following cut-points will be used for cardiovascular and metabolic parameters: dyslipidemia- lipids (cholesterol > 240 mg/L; triglycerides >500 mg/L), hypertension- systolic blood pressure > 140 mmHG or diastolic blood pressure > 90 mmHG, diabetes - fasting glucose from venous plasma fasting glucose > 126 mg/dL.
2. Medications that could affect metabolism such as cardiac drugs, thyroid, steroids, insulin, beta blockers, SSRI's, birth control pills, etc.
3. Current use of smoking/tobacco products or initiation of smoking/tobacco during the study.
4. Eating disorders as determined by screening questionnaire
5. Adherence to specialized diet regimes, vegetarian, macrobiotic, etc.
6. Food allergies, particularly lactose intolerance.
7. Treatment for psychiatric illness of chemical dependency within the previous 6 months.
8. Pregnancy or lactation.
9. Dietary intake of ≤800 mg calcium and ≤1 servings of milk per day as assessed from 3 -24 hr diet recalls (2 week-days, 1 week-end day) conducted at baseline.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Body Composition | 6 months
  Changes in body composition will be evaluated by measuring the change in percent body fat, total fat mass, and total lean mass by DEXA

SECONDARY OUTCOMES:
Blood lipids, glucose, and insulin | 6 months
  Blood samples will be collected for the purpose of measuring triglycerides, total cholesterol, HDL-cholesterol, glucose and insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, Ed.D, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States